CLINICAL TRIAL: NCT02099318
Title: Evaluation of Effort and Time Efficiency of Surgical Theater's Surgery Rehearsal Platform (SRP) for Cerebral Aneurysm Clipping Surgery
Brief Title: Surgical Theater's Surgery Rehearsal Platform
Acronym: SRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Nicholas Bambakidis, Director, Cerebrovascular and Skull Based Surgery, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 11-12-19; 14308-01-P0195-50392 (Other: 14308-01-P0195-50392)
Record Dates: First submitted 2014-03-18; First posted 2014-03-28 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Cerebral Aneurysm Unruptured; Cerebral Aneurysm Ruptured
Keywords: Rehearsal Platform
MeSH Terms: interventions — Regulatory Factor X1

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active SRP cases (Active Comparator): SRP cases: After patients have provided written informed consent, the CT and/or MRI images obtained as part of routine preoperative care will be used to construct the model that the neurosurgeons will use in the SRP. No new or additional images will be obtained as part of this study, and the SRP modeling will rely on neuroimaging conducted as part of standard preoperative assessment. For SRP cases, prior to performing surgery, surgeons will plan and rehearse patient-specific cerebral aneurysm surgery. Similarly to the CT/MRI studies, the SRP will be available for the surgeons during the surgery for evaluation of optional surgery approaches.
  Interventions: Other: Active SRP cases
- Control cases (Placebo Comparator): Control cases: The control group will be randomly selected according to a predetermined alternating sequence of consecutive prospectively video recorded aneurysm cases. Informed consent from all patients in both the control and SRP groups will be obtained.
  Interventions: Other: Control cases

INTERVENTIONS:
Other: Active SRP cases — The SRP involves preoperative rehearsal and planning. Similarly to the CT/MRI studies, the SRP will be available for surgeons during the surgery for evaluation of optional surgical approaches.
  Other Names: Trade name: Surgical Rehearsal Platform; Regulation Number: 21 CFR 892.2040; Regulation Name: Picture Archiving and Commuications System; Regulatory Class: II; Product Code: LLZ
  Arms: Active SRP cases
Other: Control cases — Control cases will consist of video recorded cases done in the exact same way as they have been performed prior to the implementation of the SRP for neurosurgery cases. Due to the alternation of cases, both the SRP and control cases will take place in the same period.
  Arms: Control cases

SUMMARY:
Objectives: The objective of this clinical study is to determine if the use of the SRP will lead to improved effort and time efficiency in cerebral aneurysm surgery. For this preliminary study, the investigators will assess key time and effort variables associated with prospectively assessed SRP neurosurgery cases in comparison with cases with no SRP rehearsal. This is a single site study with one enrolling site. This study will include a total of 40 cases 20 SRP cases and 20 control cases). SRP and control cases will be randomly selected according to a predetermined alternating sequence.

DETAILED DESCRIPTION:
Overview: This study is a blinded, multicenter, randomized study comparing key effort and time variables in 20 prospective SRP cases to these same effort and time variables in 20 video recorded control neurosurgery cases. SRP and control cases will be randomly selected according to a predetermined alternating sequence.

Effort will be assessed as the number of clipping attempts and clip evaluations, as identified by a blinded, trained rater observing video recorded SRP neurosurgical cases and control neurosurgery cases. Time will be assessed as the time that the vessel was temporarily occluded as well as total microsurgical time.

To maximize the potential effects of the SRP platform on learning, cases in the protocol will be limited to those in which the Chief Neurosurgery Resident or Cerebrovascular Fellow performs a majority of the microsurgical dissection. Their participation in this study will be that of a researcher, not of a participant.

The SRP involves preoperative rehearsal and planning. Similarly to the CT/MRI studies, the SRP will be available for surgeons during the surgery for evaluation of optional surgical approaches. Control cases will consist of video recorded cases done in the exact same way as they have been performed prior to the implementation of the SRP for neurosurgery cases. Due to the alternation of cases, both the SRP and control cases will take place in the same period. Inclusion/exclusion criteria for SRP cases and control cases will define clinically similar patient groups. Only patients who, in the opinion of their physicians, qualify for the clipping procedure will be considered for this study. The purpose of this project is to determine if simulated practice for the surgeon prior to surgery using the SRP will lead to better effort and time efficiency. Findings will be used to inform development of a larger and more rigorous trial of the SRP if the preliminary results are promising. Inclusion/exclusion criteria are as follows:

Inclusion criteria:

* Patient age >=18 years old with unruptured or ruptured cerebral aneurysm in the anterior circulation for which craniotomy and microsurgery is recommended
* Patients scheduled to undergo surgery for clipping of a cerebral aneurysm
* Able to provide written informed consent

Exclusion criteria:

* Repeat of aneurysm surgery
* Previous history of craniotomy for any reason
* Previous history of non-aneurysmal hemorrhagic stroke
* Pregnancy
* Posterior circulation
* Giant (25 mm or larger) aneurysm
* Nonsaccular aneurysm

SRP cases: After patients have provided written informed consent, the CT and/or MRI images obtained as part of routine preoperative care will be used to construct the model that the neurosurgeons will use in the SRP. No new or additional images will be obtained as part of this study, and the SRP modeling will rely on neuroimaging conducted as part of standard preoperative assessment. For SRP cases, prior to performing surgery, surgeons will plan and rehearse patient-specific cerebral aneurysm surgery. Similarly to the CT/MRI studies, the SRP will be available for the surgeons during the surgery for evaluation of optional surgery approaches.

Control cases: The control group will be randomly selected according to a predetermined alternating sequence of consecutive prospectively video recorded aneurysm cases. Informed consent from all patients in both the control and SRP groups will be obtained.

Surgical care: All surgical procedures will be done according to standard of care. Except for presurgical rehearsal, it is expected that surgical procedures between historical cases and the SRP will not differ. All care received after the surgery will be routine care.

Research procedures and measures

Prior to embarking on the proposed study, PI will assign a blinded reviewer who will review the video record of all cases from both enrolling sites. This blinded reviewer will be a fully trained neurosurgeon not otherwise affiliated with the study. The reviewer will undergo a period of training whereby he or she will review a cohort of recorded aneurysm cases (not affiliated with the current study) in consultation with the primary investigator and co-investigators until such time that agreement is reached regarding the method of evaluation of outcome measures. Following training of the blinded reviewer, the study will proceed as follows:

1. Patient recruitment utilizing inclusion/exclusion criteria, including collection of demographic and clinical patient data and aneurysm characteristics.
2. All surgeries will be videotaped consistently with current procedures. All videotaping will consist of microsurgical techniques; no subject or neurosurgery resident identifying information will be revealed.
3. Blinded evaluators will view videotapes after all surgeries have been completed and will evaluate cases using the outcome measures previously described.

Subjects

Subjects will be patients admitted for surgery for clipping of cerebral aneurysm.

Recruitment

Study Population. Two centers throughout the US will screen and identify 60 subjects with unruptured or ruptured cerebral aneurysm. Patients will be identified and recruited through site emergency departments, clinical stroke services, and direct admissions to the neurological ICUs.

Case selection

It must be acknowledged that a prospectively collected control comparison does not ensure lack of bias that will lead to group differences in neurosurgical procedures between prospectively done SRP cases and controls cases. In an effort to standardize group comparisons, the control and SRP cases will all be selected on the same time period and from the practice of the surgical PI and co-investigators. The PI and surgical co-investigator are experienced neurosurgeons who are experts in cerebral aneurysm clipping surgery. Additionally, the control cohort and SRP cohort will be obtained in a consecutive manner beginning with the implementation of the study to minimize potential selection bias and in a manner representative of the clinical practice. The investigators will also attempt to standardize the groups, including individuals that have similar clinical and demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >=18 years old with unruptured or ruptured cerebral aneurysm in the anterior circulation for which craniotomy and microsurgery is recommended
* Patients scheduled to undergo surgery for clipping of a cerebral aneurysm, per a.
* Able to provide written informed consent

Exclusion Criteria:

* Repeat of aneurysm surgery
* Previous history of craniotomy for any reason
* Previous history of non-aneurysmal hemorrhagic stroke
* Pregnancy
* Posterior circulation
* Giant (25 mm or larger) aneurysm
* Nonsaccular aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Bambakidis, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Surgical Theater Platform home page — http://www.surgicaltheater.net/

RESULTS

PARTICIPANT FLOW:
Groups:
- Active SRP Cases: SRP cases: After patients have provided written informed consent, the CT and/or MRI images obtained as part of routine preoperative care will be used to construct model that the neurosurgeons will use in the SRP. No new or additional images will be obtained as part of this study, and the SRP modeling will rely on neuroimaging conducted as part of standard preoperative assessment. For SRP cases, prior to performing surgery, surgeons will plan and rehearse patient-specific cerebral aneurysm surgery. Similarly to the CT/MRI studies, the SRP will be available for the surgeons during the surgery for evaluation of optional surgery approaches.
  Active SRP cases: The SRP involves preoperative rehearsal and planning. Similarly to the CT/MRI studies, the SRP will be available for surgeons during the surgery for evaluation of optional surgical approaches.
Period: Overall Study
Arm/Group | Active SRP Cases | Control Cases
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active SRP Cases: SRP cases: After patients have provided written informed consent, the CT and/or MRI images obtained as part of routine preoperative care will be used to construct the model that the neurosurgeons will use in the SRP. No new or additional images will be obtained as part of this study, and the SRP modeling will rely on neuroimaging conducted as part of standard preoperative assessment. For SRP cases, prior to performing surgery, surgeons will plan and rehearse patient-specific cerebral aneurysm surgery. Similarly to the CT/MRI studies, the SRP will be available for the surgeons during surgery for evaluation of optional surgery approaches.
  Active SRP cases: The SRP involves preoperative rehearsal and planning. Similarly to the CT/MRI studies, the SRP will be available for surgeons during the surgery for evaluation of optional surgical approaches.
  Inclusion criteria:
  * Patient age >=18 years old with unruptured or ruptured cerebral aneurysm in the anterior circulation f
- Total: Total of all reporting groups
Arm/Group | Active SRP Cases | Control Cases | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Number; unit: Number]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Full Range); unit: years] | 52 [32 to 72] | 52 [32 to 72] | 52 [32 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Aneurysm Clip Time
Description: Number of Clipping attempts:
  1. Applying a clip (i.e., closing a clip on the aneurysm)
  2. Removing a clip (i.e., a clip was applied on the aneurysm and then removed)
  3. Adjusting a clip (i.e., the clip was applied on the aneurysm and then opened, adjusted, and closed again).
Time Frame: At time of surgery-Time (minutes/seconds) from first clip attempt to final clip position(up to 5 minutes)
Population: Data was lost; no results can be reported
Arm/Group | Active SRP Cases | Control Cases
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Trial Aneurysm Clips Used But Not Implanted
Description: Number of Clips evaluated:
  Defined as clips that were brought in proximity to the aneurysm for evaluation (i.e., were visible in the microscopic field) but were not applied, as observed in the operating microscope's video.
Time Frame: At time of surgery-Time (minutes/seconds) from first clip to contact aneurysm to final clip placement
Population: Data was lost; no results can be reported
Arm/Group | Active SRP Cases | Control Cases
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Temporary Clip Time
Description: Total Number of minutes of temporary clip occlusion:
  Defined as the time the temporary clip is released from the clip applier until the temporary clip is removed. (For several temporary occlusions, a cumulative total of all temporary occlusions and total time of overall temporary occlusion time as observed in the operating microscope's video.)
Time Frame: At time of surgery-Total time (minutes/seconds) of all temporary clip applications to all temporary clip removal
Population: Data was lost; no results can be reported
Arm/Group | Active SRP Cases | Control Cases
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Microsurgical Time
Description: Number of minutes of total microsurgical time:
  Defined as the time elapsed from the time the aneurysm was first observed in the OR microscope until the time that the final clip was applied
Time Frame: At time of surgery-Total time (minutes/seconds) from aneurysm first seen in video to final clip placement
Population: Data was lost; no results can be reported
Arm/Group | Active SRP Cases | Control Cases
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Wasted Number of Aneurysm Clips
Description: Number of of aneurysm clips wasted according to OR records.
Time Frame: At time of surgery-Time (minutes/seconds) from first aneurysm clip attempt to final clip placement
Population: Data was lost; no results can be reported
Arm/Group | Active SRP Cases | Control Cases
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Active SRP Cases: SRP cases: After patients have provided written informed consent, the CT and/or MRI images obtained as part of routine preoperative care will be used to construct the model that the neurosurgeons will use in the SRP. No new or additional images will be obtained as part of this study, and the SRP modeling will rely on neuroimaging conducted as part of standard preoperative assessment. For SRP cases, prior to performing surgery, surgeons will plan and rehearse patient-specific cerebral aneurysm surgery. Similarly to the CT/MRI studies, SRP will be available for the surgeons during the surgery for evaluation of optional surgery approaches.
  Active SRP cases: The SRP involves preoperative rehearsal and planning. Similarly to the CT/MRI studies, the SRP will be available for surgeons during surgery for evaluation of optional surgical approaches.
  Inclusion criteria:
  * Patient age >=18 years old with unruptured or ruptured cerebral aneurysm in the anterior circulation for w
Arm/Group | Active SRP Cases | Control Cases
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No